CLINICAL TRIAL: NCT03189706
Title: Phase II Study of Hu3F8, Irinotecan/Temozolomide and Sargramostim (HITS) Chemoimmunotherapy for High-Risk Neuroblastoma
Brief Title: Study of Chemoimmunotherapy for High-Risk Neuroblastoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-251
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma (NB)
Keywords: Hu3F8; Irinotecan; Temozolomide; Sargramostim; Chemoimmunotherapy; 17-251
MeSH Terms: conditions — Neuroblastoma | interventions — Irinotecan; Temozolomide; naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: This is a pilot study of HITS in patients with resistant NB.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hu3F8, Irinotecan/Temozolomide and Sargramostim (HITS) (Experimental): Each cycle consists of four doses of hu3F8, five doses each of irinotecan and temozolomide and five doses of GM-CSF.
  Interventions: Drug: Irinotecan; Drug: temozolomide; Biological: Hu3F8; Drug: GM-CSF

INTERVENTIONS:
Drug: Irinotecan — 50mg/m^2/day IV will be administered from day 1-5
Drug: temozolomide — (given concurrently with Irinotecan) 150mg/m^2/day orally
Biological: Hu3F8 — 2.25mg/kg IV will be administered on days 2, 4, 8 and 10
Drug: GM-CSF — 250mcg/m2/day SC will be administered on days 6-10

SUMMARY:
The purpose of this study is to find out whether an experimental drug called Hu3F8 can be given with the chemotherapy drugs irinotecan and temozolomide and another drug called GM-CSF. The investigators want to find out if this combination is safe and what effect it has on the participant and the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by international criteria,.e., histopathology (confirmed by the MSK Department of Pathology) or bone marrow metastases plus high urine catecholamine levels
* High-risk NB as defined as any of the following:

  * Stage 4 with MYCN amplification (any age)
  * Stage 4 without MYCN amplification (>1.5 years of age)
  * Stage 3 with MYCN amplification (unresectable; any age)
  * Stage 4S with MYCN amplification (any age)
* Patients fulfill one of the following criteria:

  1. Have evidence of soft tissue disease OR
  2. If they only have osteomedullary disease at protocol enrollment, they should have:

     * Had previously received Hu3F8+GMCSF therapy AND have had less than a complete response to it OR
     * Had progressed progressive disease after their most recent anti-neuroblastoma therapeutic regimen
* Patients must have evaluable (microscopic marrow metastasis, elevated tumor markers, positive MIBG or PET scans) or measurable (CT, MRI) disease documented after completion of prior systemic therapy.
* Prior treatment with murine and hu3F8 is allowed.
* Prior treatment with irinotecan or temozolomide is permitted.
* Patients with prior m3F8, hu3F8, ch14.18 or hu14.18 treatment must have a negative HAHA antibody titer. Human anti-mouse antibody positivity is allowed.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Patients with CR/VGPR disease
* Existing severe major organ dysfunction, i.e., renal, cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity ≥ grade 3 except for hearing loss, alopecia, anorexia, nausea, and hypomagnesemia from TPN, which may be grade 3
* ANC < 500/uL
* Platelet count <30K/uL
* History of allergy to mouse proteins
* Active life-threatening infection
* Inability to comply with protocol requirements
* Women who are pregnant or breast-feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  The regimen will be considered safe if there are no toxicities requiring discontinuation of therapy in at least 9/10 patients during the first two cycles.
response rate (CR+PR) | 2 years
  Response assessment will be based on the best response over the course of four cycles. Disease response for NB will use the International NB Response Criteria. Patients who withdraw from the study prior to cycle 4 with < partial response will also not be considered evaluable for response and will be replaced.

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm